CLINICAL TRIAL: NCT03579121
Title: Genomic Opioid Optimization of Dosing and Selections (GOODS) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Molly B. Kraus, Assistant Professor of Anesthesiology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 17-006577
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Perioperative/Postoperative Complications
Keywords: pharmacogenomics; preoperative evaluation; perioperative opioid use
MeSH Terms: conditions — Postoperative Complications | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Intervention Model Description: All subjects meeting inclusion/exclusion criteria will undergo pharmacogenomic testing. A pharmacist will review the pharmacogemic report and make recommendations for patients in the interventional group. The anesthesiologist and orthopedic surgeon will use that information for preoperative clinical decisions related to anesthesia and analgesia.
Who Masked: Participant
Masking Description: Participants will not be aware of which arm of the study they are enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacogenomic (PGx) guided (Experimental): Subjects will have Pharmacogenomic (PGx) testing preoperatively. The pharmacists will review results and make recommendations to the anesthesia and orthopedic teams for perioperative anesthesia and analgesia. The teams will use this information to drive clinical decisions as they see fit.
  Interventions: Other: Pharmacogenomic (PGx); Other: Review results
- Control (Active Comparator): Subjects will undergo Pharmacogenomic (PGx) preoperatively but the results will be sealed until completion of treatment and clinicians will not have access to this information. These patients will undergo standard treatment dosing and medication selection.
  Interventions: Other: Pharmacogenomic (PGx)

INTERVENTIONS:
Other: Pharmacogenomic (PGx) — Administer a pharmacogenomics test (buccal swab) during the pre-operative setting
Other: Review results — Pharmacogenomic (PGx) results reviewed by the clinicians during their treatment and the results may guide clinical decisions.
  Arms: Pharmacogenomic (PGx) guided

SUMMARY:
The researchers are conducting this study to see if pharmacogenomic testing before surgery helps the doctor to choose which medications will work best for the patient.

DETAILED DESCRIPTION:
Participants, undergoing total knee replacements, will be randomized into two groups. Both groups will receive pharmacogenomics (PGx) testing preoperatively. The PGx guided group will have their results reviewed by the clinicians during their treatment and the results may guide clinical decisions. The control group results will be sealed until completion of treatment and clinicians will not have access to this information. These participants will undergo standard treatment dosing and medication selection.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary total knee arthroplasty
* Patients must understand and provide written informed consent and HIPAA authorization prior to initiation of any study-specific procedures.

Exclusion Criteria:

* Patients with a current diagnosis of chronic pain
* Patients requiring narcotics for greater than one week prior to surgery
* Patients with chronic kidney disease with a pre-op creatinine greater than 1.5
* Patient preference or need for spinal anesthesia rather than general anesthesia
* Patient planned for robotic surgical approach

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Overall Benefit of Analgesic Score (OBAS) | baseline, 48 hours following PACU discharge
  The overall benefit of analgesia score (OBAS) is a daily multi-dimensional survey that assesses analgesia benefits, opioid-related adverse events (ORAEs), and patient satisfaction. It is a seven-item scale, with items ranging from( 0 = not at all) to(4 = very much). To calculate the Total OBAS score, compute the sum of scores in items 1-6 and add '4-score in item 7'. Low score indicates high benefit.

SECONDARY OUTCOMES:
Change in prescription pattern for postoperative pain control. | baseline, 48 hours following PACU discharge
  Overall benefit of change in opioid prescription
Change in Opioid requirements | baseline, 48 hours following PACU discharge
  Opioid doses will be recorded and converted into morphine equivalents.
Changes in opioid use perioperatively based on pharmacogenomic testing | baseline, 48 hours following PACU discharge
  Opioid doses will be recorded and converted into morphine equivalents.

CONTACTS AND LOCATIONS:
Overall Officials: Molly B Kraus, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kraus MB, Bingham JS, Kekic A, Erickson C, Grilli CB, Seamans DP, Upjohn DP, Hentz JG, Clarke HD, Spangehl MJ. Does Preoperative Pharmacogenomic Testing of Patients Undergoing TKA Improve Postoperative Pain? A Randomized Trial. Clin Orthop Relat Res. 2024 Feb 1;482(2):291-300. doi: 10.1097/CORR.0000000000002767. Epub 2023 Aug 18. PMID 37594401
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials